CLINICAL TRIAL: NCT05782530
Title: Prevalence of Tattoos and Piercings in Healthcare Using the Example of Obstetrics Workers (TattOBS)
Brief Title: Prevalence of Tattoos and Piercings in Healthcare Using the Example of Obstetrics Workers
Acronym: TattOBS
Status: Withdrawn | Type: Observational
Why Stopped: No consent of the works council
Sponsor: Martin-Luther-Universität Halle-Wittenberg (Other)
Responsible Party: Principal Investigator, Marcus Riemer, MD, Principal Investigator, Martin-Luther-Universität Halle-Wittenberg
Other Study IDs: UKGEB002
Record Dates: First submitted 2023-03-10; First posted 2023-03-23 (Actual); Last update posted 2025-03-14 (Actual); Status verified 2025-03

CONDITIONS: Acceptance, Social

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- medical stuff in obstetrics: medical doctors, nurses, midwives

SUMMARY:
Tattoos and piercings as body decorations have developed into an art form over the last few decades and its social recognition is growing. However, critics also speak of an excessive lifestyle when tattooing or piercing.

The data from the questionnaires should examine how widespread tattoos and piercings are among medical staff and thus make a statement on acceptance.

ELIGIBILITY:
Inclusion Criteria:

* medical stuff in obstetrics
* minimum 18 years old

Exclusion Criteria:

* language barrier
* uncompleted questionnaire

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: medical stuff (nurses, medical doctors, midwives) working in obstetrics
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2023-04-01 (Actual); Primary Completion 2023-05-30 (Actual); Study Completion 2023-07-31 (Actual)

PRIMARY OUTCOMES:
Prevalence of tattoos and piercings in healthcare using the example of obstetrics workers | 3 months
  Measurement of self-reported tattoos and piercings by a questionnaire